CLINICAL TRIAL: NCT06111677
Title: SOFA and APACHE II Scoring Systems for Predicting Outcome of Neurological Patients Admitted in a Tertiary Hospital Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Sumit Shahi, Principal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: NeurologicalOutcomeICU
Record Dates: First submitted 2023-10-24; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to compare the discriminative power of commonly used scoring systems, namely the sequential organ failure assessment (SOFA) and acute physiology and chronic health evaluation II (APACHE II) in the intensive care unit of a tertiary care hospital.

DETAILED DESCRIPTION:
This was a retrospective cross-sectional study including patients admitted to the ICU of TU Teaching Hospital with a neurological diagnosis from January 1, 2022, to December 31, 2022. This study uses data collected prospectively as part of the Nepal Intensive Care Research Foundation (NICRF) dataset. The ICU database contained information for all components of the APACHE II and SOFA score with physiological data collected for the length of ICU, and hospital stay. Both SOFA and APACHE II were calculated from the admission data or if not available from the earliest data recorded after admission in ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with neurological diagnosis in ICUs

Exclusion Criteria:

* Patients with missing data
* Patients with ICU length of stay < 24 h

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients admitted in ICUs with neurological diagnosis from January 1, 2022 to December 31, 2022
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year
  The outcome measure was ICU mortality (survivor vs non-survivor)

CONTACTS AND LOCATIONS:
Locations (1):
- Sumit Shahi, Lalitpur, Nepal

IPD SHARING:
Plan to Share IPD: No
Individual particant data was taken from ICU database with deidentified data after taking permission